CLINICAL TRIAL: NCT00519298
Title: A Double-Blind, Placebo-Controlled, Balanced, 4-Way, Incomplete Block Design to Evaluate the Effects of a Single Administration of SAM-531 on Sleep Electroencephalogram (EEG) and Quantitative Wake EEG (qEEG) in Healthy Subjects
Brief Title: Study Evaluating Effects of SAM-531 on Sleep Electroencephalogram (EEG) and Quantitative Wake EEG in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 3193A1-1110
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Healthy; Adult
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: SAM-531
- 2 (Placebo Comparator)
  Interventions: Other: placebo
- 3 (Active Comparator)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: SAM-531 — dosage form : 0.5 mg and 5 mg capsules 3 different single doses : 1 mg, 3mg and 10 mg of SAM-531
  Arms: 1
Other: placebo — placebo
  Arms: 2
Drug: Donepezil — dosage form: 5 mg encapsulated tablets one single dose of 5 mg.
  Arms: 3

SUMMARY:
Primary: To evaluate the pharmacologic effect of single doses of SAM-531 on sleep EEG in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of non-childbearing potential aged 18 to 50 years inclusive on study day 1.
* Body mass index in the range of 18 to 30 kg/m2 and body weight greater than or equal to 50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital sign measurements, and 12-lead electrocardiogram.

Exclusion Criteria:

* Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, hematologic, neurologic, or psychiatric disease.
* Clinically significant abnormal standard EEG at screening.
* Consumption of any caffeine-containing products or alcoholic beverages within 48 hours before study day 1.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacologic effect of SAM-531 on sleep EEG in healthy subjects | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France: infomedfrance@wyeth.com
Locations (1):
- Rouffach, France